CLINICAL TRIAL: NCT05867667
Title: Cardiac Rehabilitation to Improve Breast Cancer Outcomes (CRIBCO)
Brief Title: Cardiac Rehabilitation to Improve Breast Cancer Outcomes
Acronym: CRIBCO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Budget
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2023.010; HUM00230386 (Other: University of Michigan)
Record Dates: First submitted 2023-04-27; First posted 2023-05-22 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Cardiovascular Diseases
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Rehabilitation to Improve Breast Cancer Outcomes (Experimental): 12 weeks of Cardiac Rehab
  Interventions: Other: Cardiac Rehab

INTERVENTIONS:
Other: Cardiac Rehab — Cardiac Rehab 2x per week and home exercise 1x per week: weeks 1-4 Cardiac Rehab 1x per week and home exercise 2x per week: weeks 5-8, Home exercise 3x per week: weeks 9-12

SUMMARY:
To develop a novel, proactive cardiac rehabilitation program for breast cancer survivors at enhanced risk of cardiovascular disease. Considering this program is secondary to the Michigan Medicine Cardiac Rehabilitation program's goal to manage cardiac patients, the hybrid program has been designed that limits utilization of cardiac rehabilitation to 12 visits over the first eight weeks of the intervention compared to 32 visits for cardiovascular patients.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis stage I-III
* Within 18-months of treatment completion (defined as completion of all oncologic treatments expect oral maintenance therapy)
* Age 18 years or older
* At increased risk for cardiovascular disease based on one of the following; a.Treatment with either anthracycline-based or anti-HER2 therapy-based treatment regimen plus the presence of: >2 cardiovascular heart disease risk factors (smoking, hypertension, diabetes mellitus, obesity, dyslipidemia), OR Age (>60 years) at cancer treatment, OR Left ventricular ejection fraction <50%as determined with a clinically ordered echo scan within 6 months of enrollment, b.Treatment with anthracycline followed by trastuzumab
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Planned surgery during the study period.
* Under cardiology care for known high-risk cardiovascular disease defined as the presence of any of the following: severe, unrevascularized coronary artery disease, severe valvular heart disease, advanced heart failure with a left ventricular ejection fraction <35%)
* Metastatic cancer
* Unable to exercise (e.g., inability to complete a modified stress test or musculoskeletal condition that prevents adequate participation in exercise)
* Adults unable to give consent, pregnant or lactating women, and prisoners are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular fitness (as assessed using VO2max) between baseline and after 12 weeks of participation in a tapered 12-week cardiac rehabilitation program. | up to 12 weeks after enrollment
  Change in cardiovascular fitness will be based on endpoints related to aerobic and anaerobic thresholds, including an increase in post maximal oxygen consumption (VO2max). VO2max will be assessed by indirect calorimetry (COSMED) during a graded exercise stress test using the Bruce protocol.

SECONDARY OUTCOMES:
changes in upper body strength between baseline and after a 12-week hybrid cardiac rehabilitation program. | up to 12 weeks after enrollment
  Change in muscular strength will be assessed using 5-RM tests. The tests will be performed for leg extension, leg flexion, chest press, lat pull down, and bicep curl.
changes in lower body strength between baseline and after a 12-week hybrid cardiac rehabilitation program. | up to 12 weeks after enrollment
  Change in muscular strength will be assessed using 5-RM tests. The tests will be performed for leg extension, leg flexion, chest press, lat pull down, and bicep curl.

CONTACTS AND LOCATIONS:
Overall Officials: David Lipps, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No